CLINICAL TRIAL: NCT00555100
Title: A Multicenter, Phase I Study to Determine the Maximum Tolerated Dose, Safety, Pharmacokinetics and Efficacy of Lenalidomide With and Without Dexamethasone in Japanese Subjects With Previously Treated Multiple Myeloma
Brief Title: Safety Study of Lenalidomide With and Without Dexamethasone in Japanese Subjects With Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-017
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lenalidomide — 10mg-25mg PO/day,day1-day21 of each 28day cycle. Number of Cycles:until progression or unacceptable toxicity develops.
Drug: dexamethasone — 40mg PO/day, day1-4,9-12,17-20 of each 28day cycle. Number of Cycles:until progression or unacceptable toxicity develops.

SUMMARY:
CC-5013-MM-017 is a Phase I, multicenter study to determine the maximum tolerated dose (MTD), safety profile, pharmacokinetics, and preliminary efficacy of lenalidomide with and without dexamethasone in Japanese subjects with previously treated MM. The study will consist of two cohorts: 1) Monotherapy "Maximum Tolerated Dose (MTD) Determination" Cohort; and 2) "Combination Treatment" Cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with previously treated multiple myeloma
* Measurable levels of m-protein in serum >= 0.5 g/dL [5g/L]) or urine (>= 0.2 g excreted in a 24-hour collection sample)
* ECOG performance status of 0 - 2
* Willing to follow pregnancy precautions

Exclusion Criteria:

* Patients with acute an myocardial infarction (MI) within the past 6 months, or patients with a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the past 3 years
* Patients with tuberculous diseases, herpes simplex keratitis, systemic mycosis or other active infectious diseases
* Patients with non-controlled diabetes, hypertension, digestive ulcer or glaucoma
* Patients with posterior subcapsular cataracts
* Patients with mental illness
* Patients with past histories or complications which make the Investigator or other staff member deem them inappropriate for this study
* Pregnant or lactating females
* Grade 2 or worse neuropathy
* Any of the following laboratory abnormalities:

Absolute neutrophil count (ANC) < 1,000cells/mL Platelet count < 75,000/mL Serum creatinine > 2.5 mg/dL Serum SGOT/AST or SGPT/ALT > 3.0 x upper limit of normal (ULN)

* Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for >= 3 years. - Patients who received radiation therapy within 14 days of the start of study drug
* Patients with scars from a recent viscus operation
* Patients with history of a desquamating (blistering) rash while taking thalidomide
* Patients with prior use of lenalidomide
* Patients with known HIV positivity.
* Patients who used cytotoxic chemotherapeutic agents, immunomodulating agents, or other experimental agents (agents that are not commercially available) intended for the treatment of MM within 28 days of the start of lenalidomide therapy.
* Patients with known history of hypersensitivity to dexamethasone.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07-01 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2010-12-01 (Actual)

PRIMARY OUTCOMES:
DLT | first cycle (28 days)

SECONDARY OUTCOMES:
Efficacy (M-protein) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Masaaki Takatoku, M.D., Study Director — Celgene K.K.
Locations (5):
- Japan (5):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Niigata Cancer Center Hospital, Niigata
  - Keio University Hospital, Tokyo

REFERENCES:
- [Background] Iida S, Chou T, Okamoto S, Nagai H, Hatake K, Murakami H, Takagi T, Shimizu K, Lau H, Takeshita K, Takatoku M, Hotta T. Lenalidomide plus dexamethasone treatment in Japanese patients with relapsed/refractory multiple myeloma. Int J Hematol. 2010 Jul;92(1):118-26. doi: 10.1007/s12185-010-0624-7. Epub 2010 Jun 18. PMID 20559759